CLINICAL TRIAL: NCT06275646
Title: Comparison Of Outcome Of Autologus Platelet Rich Plasma Membrane Plus Dartos Flap Versus Simple Dartos Flap In Hypospadias Surgery
Brief Title: Comparison Of Outcome Of Different Layers in Hypospadias Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children Hospital and Institute of Child Health, Lahore (Other)
Responsible Party: Principal Investigator, Muhammad Adeel Ashiq, Principal Investigator, Children Hospital and Institute of Child Health, Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Adeel2
Record Dates: First submitted 2024-02-12; First posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Hypospadias
Keywords: Hypospadias; platelet rich plasma; distal penile hypospadias
MeSH Terms: conditions — Hypospadias

STUDY DESIGN:
Intervention Model Description: randomized control trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A dartos flap and PRP layer (Experimental): dartos flap and PRP layer was applied in hypospadias surgery as additional layer
  Interventions: Other: PRP layer; Other: dartos flap
- preputial dartos flap layer (Experimental): preputial dartos flap layer applied as additional layer
  Interventions: Other: dartos flap

INTERVENTIONS:
Other: PRP layer — platelet rich plasma layer was applied in addition to dartos flap
  Arms: A dartos flap and PRP layer
Other: dartos flap — dartos flap alone was used

SUMMARY:
To compare the outcome of applying autologous platelet-rich plasma membrane layer and dartos fascial flap versus only dartos fascial flap in mid and distal penile hypospadias surgery. A total of 220 patients fulfilling the selection criteria were admitted after taking informed consent. Cases were randomly divided into groups A and B using a random generator of the Excel program. In group A, dartos flap and PRP sheet layer were applied and in group B, only a preputial dartos fascial flap was applied

DETAILED DESCRIPTION:
Objective To compare the outcome of application of autologous platelet-rich plasma membrane layer and dartos fascial flap versus only dartos fascial flap in mid and distal penile hypospadias surgery.

Methods This randomized controlled trial was conducted at Pediatric General surgical department, the Children's hospital and the University of Child health, Lahore for the period of 12 months. Non probability, purposive sampling was used for data collection and randomization was done to assign the treatment. Total of 220 patients fulfilling the selection criteria were admitted after taking an informed consent. Cases were randomly divided into two groups A and B using random generator of Excel program. In group-A, dartos flap and PRP sheet layer was applied and in group-B, only a preputial dartos fascial flap was applied.

ELIGIBILITY:
Inclusion Criteria:

* patients (Age 6months to12 years) with mid, distal penile or sub coronal hypospadias having minimal chordae were included in the study

Exclusion Criteria:

* Patients having proximal hypospadias, moderate to severe chordae, previously operated cases, a preoperative androgens treatment (for example in penoscrotal hypospadias and small sized phallus) were excluded from study

Ages: 6 Months to 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — only males with hypospadias
Enrollment: 220 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
wound infectiom | 30 days
  local wound infection assessed by southampton wound assessment scale where 0 means excellent and 4 means worst
frequency of glans dehiscence | 30 days
  glans dehiscence observed
frequency of meatal stenosis | 30 days
  meatal stenosis assessed on examination

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Adeel Ashiq, M.S, Principal Investigator — CHUCHS
Locations (1):
- The Children Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No